CLINICAL TRIAL: NCT05567003
Title: Percutaneous Endoscopic Laser Incision for Benign Biliary Strictures: Prospective Evaluation of Safety and Efficacy
Brief Title: Percutaneous Endoluminal Benign Biliary Laser
Acronym: PEBBL
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study did not meet enrollment targets.
Sponsor: University of California, Los Angeles (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Ravi N. Srinivasa, MD, Professor of Vascular and Interventional Radiology, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-001910
Record Dates: First submitted 2022-09-30; First posted 2022-10-05 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Benign Biliary Strictures With Current or Prior Biliary Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with benign biliary strictures (Other): Patients with benign biliary strictures with current or prior biliary obstruction, who would otherwise receive standard treatment with long-term biliary tube drainage.
  Interventions: Procedure: Percutaneous transhepatic cholangioscopic (PTCS) laser incision

INTERVENTIONS:
Procedure: Percutaneous transhepatic cholangioscopic (PTCS) laser incision — Infrared percutaneous transhepatic cholangioscopic guided holmium laser incision for treatment of benign biliary strictures.

SUMMARY:
This study is being done to evaluate the safety and efficacy of Percutaneous transhepatic cholangioscopic (PTCS) laser incision as an ancillary therapy to traditional approaches such as balloon dilation and large drain placement for Benign Biliary Strictures (BBS).

Narrowing or blockage of the bile ducts (biliary stricture) is a difficult to treat medical condition that leads to life-threatening complications. Treatment usually involves multiple procedures or surgeries spanned over months or years, and in many cases, leads to the need for a life-long tube that drains bile fluid outside of the body and into a bag. PTCS laser incision is a promising new treatment for bile duct strictures. The procedure is performed by an Interventional Radiologist who uses a tiny camera (endoscope) and a laser through a small hole in the skin to open up the blocked or narrowed duct. This allows bile to flow freely where it is supposed to go (without a tube) so that it does not backup up and cause life-threatening problems. Based on early experience from patients who have had this procedure done, it appears to be safe and effective, and may lead to needing fewer procedures over time, with the possibility of living without a tube or drain. The main goal of this study is to confirm the safety and efficacy of PTCS laser incision in a series of patients with benign biliary strictures who would otherwise receive standard treatment with long-term biliary tube drainage.

DETAILED DESCRIPTION:
PTCS-guided holmium laser incision is a promising new adjuvant treatment for benign biliary strictures. Real-time monitoring under direct endoscopic visualization provides an invaluable opportunity for Interventional Radiologists to safely perform targeted diagnosis and treatment within the biliary system. Despite limited literature on the subject, there are several potential advantages of bringing cholangioscopic laser incision to the Interventional Radiology (IR) suite.

First, management of biliary strictures and their sequelae is commonplace in daily IR practice. With increasing sophistication of modern therapeutics including ablation, lithotripter, stent and retrieval devices, there is increasing risk to using fluoroscopy alone to perform complex interventions in a three-dimensional space. Endoscopy allows real-time monitoring of treatment progress and potential complications. For example, an operator using fluoroscopy could not identify iatrogenic haemobilia as readily as an operator using endoscopy, and delayed recognition of such a complication could have lethal consequences. Fortunately, hemorrhagic complications encountered in the IR suite can be treated by trans-arterial embolization. Endoscopic visualization also allows an operator to more precisely characterize the etiology, extent, and other specific features of a focal narrowing within the bile ducts, thus facilitating a more targeted and patient-specific approach to diagnosis and treatment. Conversely, a filling defect seen on conventional cholangiography is nonspecific and can result in an indeterminant biopsy or lead to inappropriate treatment.

Second, PTCS-guided laser incision can improve clinical outcomes and potentially be a definitive treatment option for patients with recalcitrant BBS who otherwise require life-long percutaneous drainage. Unlike mechanical dilation techniques such as balloon cholangioplasty and stenting, the holmium laser addresses the root cause of stricture by incising excess fibrotic intraluminal tissue and restoring patency to the native bile duct, while also eliminating the need for an indwelling device that can become a nidus for infection. In contrast to radiofrequency (RF) ablation or the neodymium laser, the holmium laser's short depth of penetration and selective wavelength for water absorption results in precise tissue dissection by way of vaporization, with minimal thermal damage to surrounding tissues. This results in less inflammation and trauma to the bile ducts, which are the major culprits of re-stenosis. Additionally, the device can be employed simultaneously for lithotripsy of concomitant biliary stones which must be removed at the time of intervention to prevent cholangitis and stricture recurrence.

Third, PTCS-guided laser incision has the potential to reduce patient morbidity and improve quality of life. By decreasing the total number of interventions and amount of time patients require a drainage catheter or other indwelling device, a decrease in cumulative procedural and stricture-related complications would likewise be expected. In contrast to 1 or 2 PTCS sessions, standard protocols involve multiple interventions over the course of several months, during which time patients are expected to self-manage a biliary drainage bag and continuously monitor for signs and symptoms of cholangitis and elevated bilirubin. Following a capping trial, still some 20-30% of patients develop recurrent stricture, many of whom have no other option but to continue indefinitely with a drainage tube while carrying a life-long risk of recurrent cholangitis and other obstructive phenomena. The improved efficiency of PTCS-guided laser incision also implicates a potential to decrease procedure-related costs, use of hospital and departmental resources, and radiation exposure to patients. In the past, the high overhead cost of reusable endoscopes prohibited most IR groups from adopting endoscopy. However, the development of new disposable low-profile devices has eliminated the financial barrier to entry for IR-operated endoscopy and may yield cost savings over time with less angiography suite usage.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of Benign Biliary Strictures (BBS)
2. Clinical and/or laboratory evidence of biliary obstruction (current or prior)
3. Age 18 years or older at the time of intervention

Exclusion Criteria:

1. Patients with a diagnosis of malignant biliary stricture at the time of enrollment
2. Patients who are subsequently diagnosed with malignant biliary stricture during the study period
3. Liver transplantation within the last 90 days
4. Active cholangitis or sepsis
5. Emergent need for biliary decompression
6. Patients with a diagnosis of primary sclerosing cholangitis with presence of 3 or more strictured segments
7. Patients with a life-expectancy of less than 36 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Post Procedure Adverse Events | Up to 24 months
  Safety evaluated by cumulative rates of post-interventional complications after PTCS-guided laser incision.
  1. Complications will be reported according to the Society of Interventional Radiology Adverse Event (AE) classification system.
  2. Safety will be reported as 30-day composite of all post-procedure AEs.
  3. Complications will be further qualified and quantified by AE severity category and individual AE types.
Feasibility of Procedure | Up to 24 months
  Feasibility evaluated by technical success of PTCS-guided laser incision.
  a. Technical success defined as endoscopic and cholangiographic evidence of improved patency at the time of intervention.

SECONDARY OUTCOMES:
Primary Bile Duct Patency | Up to 24 months
  Primary bile duct patency evaluated as mean time to first stricture recurrence.
  1. Stricture recurrence will be defined as clinical and/or radiographic evidence of biliary occlusion requiring additional therapy.
  2. The date of PTCS or post-intervention biliary catheter removal will mark the time of initiation.
Tube-Free Survival | Up to 12 months
  Tube-free survival evaluated as cumulative time survived without a biliary device during the study period.
  1. Duration of time that patients require a biliary catheter or stent during follow-up period will be subtracted from the 12-month total.
  2. If a device is subsequently removed, tube-free survival time will continue to be accrued up to 12 months post-treatment.
12-Month Cumulative Complications | Up to 12 months
  12-month cumulative complications from laser treatment or recurrent biliary disease.
  a. Composite of all PTCS- and stricture-related AEs during the 12-month follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi N Srinivasa, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No